CLINICAL TRIAL: NCT03089983
Title: Addiction, HIV and Tuberculosis in Malaysian Criminal Justice Settings
Acronym: HARAPAN II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: University of Malaya (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2000020053; 1R01DA041271 (NIH)
Record Dates: First submitted 2017-02-16; First posted 2017-03-24 (Actual); Results first posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Opioid Dependence; Addiction; HIV/AIDS; Tuberculosis; Hepatitis
Keywords: prison
MeSH Terms: conditions — Opioid-Related Disorders; Behavior, Addictive; Acquired Immunodeficiency Syndrome; Tuberculosis; Hepatitis | interventions — Isoniazid; rifapentine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Isoniazid (INH) for 26 weeks (Active Comparator): Participants will be randomized to receive INH, the standard of care in Malaysia, for 26 weeks while in prison as TB preventative treatment
  Interventions: Drug: Isoniazid
- Short-course isoniazid + rifapentine (INH + RIF) for 12 weeks (Experimental): Participants will be randomized to receive INH + RIF as TB preventative treatment for 12 weeks while in prison.
  Interventions: Drug: Isoniazid; Drug: Rifapentine

INTERVENTIONS:
Drug: Isoniazid — Participants will be randomized to receive standard INH as TB preventative treatment
Drug: Rifapentine — Participants will be randomized to receive short course INH + RIF as TB preventative treatment
  Arms: Short-course isoniazid + rifapentine (INH + RIF) for 12 weeks

SUMMARY:
The purpose of this study is to conduct empiric studies of tuberculosis (TB) among people in prison with and without a history of opioid dependence. A RCT of latent TB infection prevention strategies among HIV+ and HIV- prisoners with high prevalence of hepatitis C (HCV) using standard 40-week daily isoniazid (40H) vs short-course weekly isoniazid + rifapentine (12HR). Investigators will also use this data, and publicly available data to complete agent-based modeling for comparative and cost-effectiveness of various TB screening and treatment strategies among prisoners.

DETAILED DESCRIPTION:
Screening: All newly admitted prisoners (80-120 new inmates on admission days) undergo a complete assessment, including a brief exam and mandatory rapid HIV test by the prison medical unit. Each prisoner waiting to be evaluated will be invited for participation in TB screening activities (not currently part of standard care). If they verbally assent to wanting to learn more in a group session, their names and ID will be recorded and then invited for informed consent privately, followed by a brief survey, WHO symptom assessment, tuberculin skin testing (TST) with reading after 72 hours, sputum induction on 2 consecutive mornings for AFB smear, TB culture (results back 6-8 weeks using the BACTEC MGIT 960 liquid culture gold standard), and point-of care (POC) Gene Xpert. Each person will have phlebotomy for HBV and HCV Ab, LFTs, and if HIV+, CD4 testing (all of these are POC using Alere™). For those with CD4<50, they will undergo POC low-cost, urinary TB-LAM lateral flow testing (sensitivity=67%) (Alere™ Determine) to identify disseminated TB. Additional demographic, drug use, and TB risks will also be assessed along with prison data (release date, previous incarcerations, type of offense). Participants will then undergo CXR testing. A TB specialist will review all patients and results, ensuring that patients with suspected TB initiate treatment. All suspected or confirmed cases active TB cases in HIV+ prisoners will have ART initiated after 2 weeks of TB treatment initiation (if CNS TB not suspected) if CD4<50 and within 8 weeks for all others.

Trial: All HIV+ and HIV- prisoners with latent TB infection (LTBI) (TST reaction 10 mm or greater) from screening will be asked to participate in the trial. Enrolled participants will undergo block stratified randomization, stratifying on three factors: a) CD4<350; b) HCV Ab status; and c) ART status. After randomization and allocation to 12HR or 40H, participants will be provided 12HR weekly (12 weeks) and INH daily (26 weeks) as directly observed therapy. Every 4 weeks, patients will be monitored for AST/ALT and adverse side effects. Premature treatment discontinuation will occur for any DAIDS Grade 4 toxicity or patient refusal to continue.

The focus of this registration is the RCT. Outcomes measures were updated to match most recent protocol March 2025.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria (screening):

* Age ≥ 18 years
* Newly admitted inmate at Kajang Prison

Inclusion Criteria (Trial):

* Age ≥ 18 years HIV-1 seropositivity
* Confirmed LTBI (TST ≥ 5mm if HIV+; TST ≥ 10 mm if HIV-)
* Meets DSM-V criteria for opioid dependence
* >9 months before release (to ensure treatment completion in prison)
* AST/ALT < 3x upper limit normal

Exclusion Criteria:

* Unable to provide informed consent
* On a protease inhibitor
* Women who are pregnant or are planning on becoming pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Altice, MD, Principal Investigator — Yale University; Adeeba Kamarulzaman, MBBS, Principal Investigator — University of Malaya; Sheela Shenoi, MD, Principal Investigator — Yale University
Locations (1):
- Kajang Prison, Kajang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 327 eligible participants, 316 participants consented, 4 participants were excluded prior to randomization, and 312 randomized
Period: Overall Study
Arm/Group | Standard Isoniazid (INH) for 26 Weeks | Short-course Isoniazid + Rifapentine (INH + RIF) for 12 Weeks
Started | 156 | 156
Initiated Treatment | 152 | 153
Completed | 114 | 127
Not Completed | 42 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Isoniazid (INH) for 26 Weeks | Short-course Isoniazid + Rifapentine (INH + RIF) for 12 Weeks | Total
Number analyzed (Participants) | 156 | 156 | 312
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 43 [37 to 49] | 42 [35 to 49] | 42.5 [37 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 156 | 156 | 312
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Malay | 104 | 95 | 199
  Chinese | 17 | 17 | 34
  Indian | 34 | 39 | 73
  Other | 1 | 5 | 6
Region of Enrollment [Number; unit: participants]
  Malaysia | 156 | 156 | 312
Education level [Count of Participants; unit: Participants]
  Primary school and below | 31 | 52 | 83
  secondary school | 119 | 100 | 219
  Tertiary school | 6 | 4 | 10
Marital Status [Count of Participants; unit: Participants]
  Single/partner | 91 | 89 | 180
  Married | 44 | 33 | 77
  Widowed/Divorced | 21 | 34 | 55
Employed prior to incarceration [Count of Participants; unit: Participants] | 136 | 119 | 255
Previously incarcerated [Count of Participants; unit: Participants] | 144 | 150 | 294
Median number of prior incarcerations [Median (Inter-Quartile Range); unit: incarcerations] | 9 [5 to 15] | 9 [5 to 15.25] | 9 [5 to 15]
Homelessness [Count of Participants; unit: Participants] | 24 | 28 | 52
Previous TB disease [Count of Participants; unit: Participants] | 10 | 10 | 20
Previous diagnosis of HIV [Count of Participants; unit: Participants] | 22 | 17 | 39
Number of Participants previously prescribed ART [Count of Participants; unit: Participants] | 17 | 9 | 26
Previously taking ART prior to prison entry [Count of Participants; unit: Participants] | 12 | 6 | 18
Total people with HIV [Count of Participants; unit: Participants] | 23 | 18 | 41
Previous Opioid Use [Count of Participants; unit: Participants] | 124 | 130 | 254
Positive Rapid Opioid Dependence Screen (RODS) (≥3) on enrollment [Count of Participants; unit: Participants] — Screening tool to assess opioid dependence and the need for services for opioid use or withdrawal that require medical attention. A diagnosis of opioid dependence is made if three or more affirmative responses are given.
  Participants | 112 | 124 | 236
Previous intravenous drug use (IVDU) [Count of Participants; unit: Participants] | 67 | 67 | 134
Elevated (>4) Alcohol Use Disorders Identification Test (AUDIT) C score [Count of Participants; unit: Participants] — The possible AUDIT-C scores range from 0 to 12 with higher scores suggesting potential alcohol problems.
  Participants | 18 | 18 | 36
Median days since prison entry [Median (Inter-Quartile Range); unit: days] | 67 [53 to 108.5] | 76.5 [56 to 149.5] | 71 [55 to 127]
Positive Hepatitis C [Count of Participants; unit: Participants] | 69 | 70 | 139
Median Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m²] | 22.6 [20.74 to 24.33] | 21.51 [19.57 to 24.07] | 22.2 [20.23 to 24.17]

OUTCOME MEASURES:

1. Primary Outcome: TB Treatment Completion Rates in Prison
Description: TB treatment completion in prison will be verified using medical records. All TB treatment in prison will be administered under directly observed therapy (DOTs), and treatment administration will be recorded in the participant's prison medical record. Data presented here is the number of participants that completed TB treatment of those that initiated treatment.
Time Frame: 3 to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Isoniazid (INH) for 26 Weeks | Short-course Isoniazid + Rifapentine (INH + RIF) for 12 Weeks
Number analyzed (Participants) | 152 | 153
Participants | 114 | 127
Statistical Analysis 1: Comparison: Standard Isoniazid (INH) for 26 Weeks vs Short-course Isoniazid + Rifapentine (INH + RIF) for 12 Weeks; Test type: Superiority; p = 0.08, t-test, 2 sided

2. Secondary Outcome: TB Treatment Adherence
Description: TB treatment adherence in prison will be verified using medical records. All TB treatment in prison will be administered under directly observed therapy (DOTs), and treatment administration will be recorded in the participant's prison medical record. Data presented here is the number of participants that adhered to TB treatment of those that initiated treatment.
Time Frame: monthly for up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Isoniazid (INH) for 26 Weeks | Short-course Isoniazid + Rifapentine (INH + RIF) for 12 Weeks
Number analyzed (Participants) | 152 | 153
Participants | 9 | 117

3. Secondary Outcome: Discontinuation Due to Experiencing an Adverse Event
Description: The number of participants that discontinued the trial due to experiencing an Adverse Event
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Isoniazid (INH) for 26 Weeks | Short-course Isoniazid + Rifapentine (INH + RIF) for 12 Weeks
Number analyzed (Participants) | 156 | 156
Participants | 10 | 1

4. Secondary Outcome: Acceptability of Starting the Trial
Description: Acceptability defined as the number of eligible participants that agreed to consent
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Participants: Eligible participants post screening.
Arm/Group | Eligible Participants
Number analyzed (Participants) | 327
Participants | 316

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Short-course Isoniazid + Rifapentine (INH + RIF) for 12 Weks: Participants will be randomized to receive INH + RIF as TB preventative treatment for 12 weeks while in prison.
Arm/Group | Standard Isoniazid (INH) for 26 Weeks | Short-course Isoniazid + Rifapentine (INH + RIF) for 12 Weks
All-Cause Mortality (participants affected / at risk) | 0/156 | 0/156
Serious Adverse Events (participants affected / at risk) | 0/156 | 0/156
Other Adverse Events (participants affected / at risk) | 112/156 | 84/156
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Isoniazid (INH) for 26 Weeks (N=156) | Short-course Isoniazid + Rifapentine (INH + RIF) for 12 Weks (N=156)
Clumsiness or unsteadiness (Nervous system disorders) | 2 | 0
Dark urine (Renal and urinary disorders) | 5 | 10
Loss of appetite (Metabolism and nutrition disorders) | 13 | 5
Nausea (Gastrointestinal disorders) | 4 | 5
Vomiting (Gastrointestinal disorders) | 2 | 3
Diarrhea (Gastrointestinal disorders) | 13 | 4
Stomach pain (Gastrointestinal disorders) | 14 | 7
Yellow eyes or skin (General disorders) | 0 | 1
Blurred vision or loss of vision (Eye disorders) | 6 | 3
Fever and sore throat (Infections and infestations) | 8 | 7
Joint pain (Musculoskeletal and connective tissue disorders) | 47 | 28
Mental depression (Psychiatric disorders) | 3 | 2
Mood or other mental changes (Psychiatric disorders) | 6 | 6
Skin rashes (Skin and subcutaneous tissue disorders) | 59 | 34
Unusual bleeding or bruising (Injury, poisoning and procedural complications) | 6 | 0
Numbness, tingling, burning, or pain in hands and feet (Nervous system disorders) | 18 | 10
Unusual tiredness or weakness (General disorders) | 10 | 5
Red, orange, or brown discoloration of skin or body fluids (General disorders) | 2 | 11
Other (General disorders) | 9 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT03089983/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/83/NCT03089983/ICF_001.pdf